CLINICAL TRIAL: NCT02540343
Title: Intercultural Adaptation and Validation of the "Orebro Musculoskeletal Pain Questionnaire"-Translation and Validation of a Questionnaire
Brief Title: Intercultural Adaptation and Validation of the "Orebro Musculoskeletal Pain Questionnaire"
Acronym: Orebro-G
Status: Completed | Type: Observational
Sponsor: Balgrist University Hospital (Other)
Collaborators: Maastricht University (Other)
Responsible Party: Principal Investigator, Swanenburg, PhD, Balgrist University Hospital
Other Study IDs: Balgrist 2013-0394
Record Dates: First submitted 2015-08-21; First posted 2015-09-03 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Neck Pain
Keywords: Translation; Validation; Orebro-G
MeSH Terms: conditions — Neck Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- acute neck pain patients: Participant recently received the diagnosis of neck pain (< 30 days) >18 years old able to speak, read and write German, questionnaires
  Interventions: Other: questionnaires
- chronic neck apin patients: Participant has neck pain for a longer period of time (> 90 days) > 18 years old able to speak, read and write German, questionnaires
  Interventions: Other: questionnaires
- test persons: no neck pain > 18 years old able to speak, read and write German, questionnaires
  Interventions: Other: questionnaires

INTERVENTIONS:
Other: questionnaires — fill out all questionnaires twice

SUMMARY:
The aim of this study is to adapt and translate the Orebro Musculoskeletal Pain Questionnaire into German.

DETAILED DESCRIPTION:
Participants will fill out all questionnaires at baseline and again after three days. If the questionnaires have not been returned by day four the participant receives a reminder telephone call. Patients that do not return the questionnaires by day seven are dismissed. The baseline measurement is done at the practice the second measurement will be done by the patient at home. To send the questionnaire back the participant receives a prepaid envelope.

ELIGIBILITY:
Inclusion Criteria:

Acute:

* Recently diagnosed with neck pain (< 30 days)
* Must be able to speak, read and write German

Chronic:

* Neck problems for a longer period of time (> 90 days)
* Must be able to speak, read and write German

Healthy volunteers:

* No neck pain
* Must be able to speak, read and write German

Exclusion Criteria:

* Does not speak, read and write German
* "Red Flags" e.g. acute trauma
* Medical knowledge

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Acute and chronic neck pain patients Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2014-11; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Pain, on the German Version of the Orebro Musculoskeletal Pain Screening Questionnaire | For every patient the average study length is one week.
  Participants are asked to fill out the questionnaire twice. At the start and three to seven days after the first time.

SECONDARY OUTCOMES:
Disability, on the Neck Disability Index (NDI-G) | For every patient the average study length is one week.
  Participants are asked to fill out the questionnaire twice. At the start and three to seven days after the first time.
Pain, on Visual Analogue Pain Rating Scale (VAS) | For every patient the average study length is one week.
  Participants are asked to fill out the questionnaire twice. At the start and three to seven days after the first time.

OTHER OUTCOMES:
Voice Handicap, on the Voice Handicap Index (VHI-9) | For every patient the average study length is one week.
  Participants are asked to fill out the questionnaire twice. At the start and three to seven days after the first time.
Movement restriction, on self-reported measurements of the Range of motion of the cervical spine | For every patient the average study length is one week.
  Participants are asked to fill out the questionnaire twice. At the start and three to seven days after the first time.

CONTACTS AND LOCATIONS:
Overall Officials: Jaap Swanenburg, PhD, Principal Investigator — Balgrist University Hospital
Locations (1):
- Balgrist University Hospital, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Langenfeld A, Bastiaenen C, Brunner F, Swanenburg J. Validation of the Orebro musculoskeletal pain screening questionnaire in patients with chronic neck pain. BMC Res Notes. 2018 Mar 2;11(1):161. doi: 10.1186/s13104-018-3269-x. PMID 29499753